CLINICAL TRIAL: NCT02923076
Title: A Prospective Clinical Research Protocol of Allogeneic CCR5 delta32/delta32 Cord Blood Cell Transplantation to Cure HIV Infection
Brief Title: HIV Eradication Through Cord-blood Transplantation
Acronym: HIVECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Fundación Mutua Madrileña (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Rafael F. Duarte, Head of the Hematopietic Cell Transplantation program, Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIVECT-1501
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: HIV
Keywords: Allogeneic Hematopoietic Cell Transplantation

ARMS (1):
- Study treatment (Experimental): Allogeneic transplantation with CCR5 delta32/delta32 hematopoietic cells from cord blood.
  Interventions: Other: CCR5 delta32/delta32 cord blood transplantation

INTERVENTIONS:
Other: CCR5 delta32/delta32 cord blood transplantation

SUMMARY:
Allogeneic hematopoietic cell transplantation from a CCR5 Δ32/Δ32 unrelated donor, performed for the first time in the "Berlin patient", provides the only evidence to date of long-term control of HIV infection. Stringent criteria to select human leukocyte antigen (HLA)-matched conventional donors and low prevalence of the CCR5 Δ32/Δ32 homozygous genotype (<1%) made the pursuit of "patient number 2" unsuccessful for many years. Cord blood (CB) transplantation allows more permissive HLA-matching criteria, making the search for HLA-compatible Δ32/Δ32 CB units potentially feasible for transplantation of HIV-infected individuals.

The investigator team involved in this trial has recently reported the first such case of CCR5 delta32/delta32 CB transplantation in a patient with HIV infection, showing a reduction of the patient's latent viral reservoir and, upon achievement of full CB chimerism, resistance of his CD4 T-lymphocytes to infection by HIV. This proof of concept led the Spanish National Transplant Organization (ONT) to generate an inventory of over 150 CCR5 Δ32/Δ32 CB units readily available for transplant.

From this initial evidence and repository of CB units, financial support from the Fundación Mutua Madrileña (FMM) has allowed the investigators to launch this first pilot clinical trial in this indication. The study was launched in January 2016 at Hospital Universitario Puerta de Hierro Majadahonda. All HIV virology and reservoir analyses are carried out by the AIDS Immunopathology Unit at the Spanish Instituto de Salud Carlos III. Three additional transplant centres in Spain will also shortly open the trial.

ELIGIBILITY:
Inclusion Criteria:

* Inform consent, that will be previously approved by the board, is required in order to carry out any procedure related to the study.
* HIV infection.
* Hematologic malignancies or any other condition with a standard indication for allogeneic hematopoietic cell transplantation. See indications by the European Society for Blood and Marrow Transplantation (EBMT). [Sureda A. et al. Indications for allo- and auto-SCT for haematological diseases, solid tumours and immune disorders: current practice in Europe, 2015. Bone Marrow Transplantation (2015) 50, 1037-1056.]
* Lack of HLA-identical related donor
* Availability of at least one cord blood unit CCR5 delta32 homozygous that meets quality standards.

Exclusion Criteria:

* Availability of HLA-identical related donor
* Contraindication for allogeneic stem cell transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
HIV infection and viral reservoir - Cell-associated total HIV-1 DNA in CD4 T cells from peripheral blood and from gut-associated lymphoid tissue (GALT): Expressed in copies per million cells. | Between 6-12 months: following discontinuation of antiretroviral therapy upon full CCR5 delta32/delta32 cord blood chimerism
HIV infection and viral reservoir - Viral copies in plasma and culture supernatants by Single Copy Assay and COBAS AMPLICOR HIV-1 Monitor v.1.5: Expressed in copies per mL. | Between 6-12 months: following discontinuation of antiretroviral therapy upon full CCR5 delta32/delta32 cord blood chimerism
Ex vivo HIV-1 infection tests on CCR5 d32/d32-derived recipients CD4 T cells - Using patient's primary isolates and laboratory strains of HIV-1 with CCR5 and CXCR4 tropism: Expressed in ng/mL of p24 ELISA. | Between 6-12 months: following discontinuation of antiretroviral therapy upon full CCR5 delta32/delta32 cord blood chimerism

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Duarte Palomino, Principal Investigator — Hospital Universitario Puerta de Hierro- Majadahonda
Locations (1):
- Hospital Universitario Puerta de Hierro- Majadahonda, Majadahonda, Madrid, Spain